CLINICAL TRIAL: NCT02118207
Title: The Impact of Predive Exercise on Repetitive SCUBA Diving
Brief Title: Exercise and Repetitive Diving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Zeljko Dujic, Professor Zeljko Dujic MD, PhD, Director of Department of Physiology, University of Split
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 264816-02
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Decompression Sickness; Endothelial Dysfunction; Neutrophil Activation; Venous Gas Emboli
Keywords: SCUBA diving; Exercise; Microparticles; Repetitive diving; Endothelial function
MeSH Terms: conditions — Decompression Sickness; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control dives 1st (Experimental): Subjects in this group complete the first 3 dives as control dives and the second 3 dives preceded by aerobic exercise
  Interventions: Other: Aerobic running exercise
- Predive exercise 1st (Experimental): Subjects complete the first 3 dives preceded by the intervention of aerobic exercise and the second 3 with no exercise as control dives
  Interventions: Other: Aerobic running exercise

INTERVENTIONS:
Other: Aerobic running exercise — 60 min of aerobic intervals completed prior to SCUBA diving

SUMMARY:
SCUBA diving frequently involves repetitive exposures over multiple days. The goal of this study was to see how exercise impacts microparticles (MPs), endothelial function, and venous gas emboli (VGE) over a series of dives.

16 divers in 2 groups each completed 6 dives. One group completed 3 control dives followed by 5 days rest then 3 dives preceded by exercise. The other group completed the opposite protocol. Flow-mediated dilation (FMD) data and blood for MP analysis was collected before and after each dive. VGE were monitored via transthoracic echocardiography 30, 60, and 90 min after surfacing. Exercise before diving consisted of 60 min running outdoors including 8x4 min intervals at 90% VO2max effort.

ELIGIBILITY:
Inclusion Criteria:

* Certified SCUBA diver
* Certified to dive by experienced Medical evaluator
* Must be able to run continuously for 45 min

Exclusion Criteria:

* Prior diagnosis of decompression sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in circulating microparticle counts | 2 weeks
  Change in circulating microparticle counts measured pre and post SCUBA diving following 6 dives spaced over 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Zeljko Dujic, MD, PhD, Principal Investigator — University of Split, School of Medicine
Locations (2):
- University of Maryland, Baltimore, Maryland, United States
- University of Split School of Medicine, Split, Croatia